CLINICAL TRIAL: NCT06509022
Title: China Cancer Foundation Beijing Hope Marathon Fund
Brief Title: Longitudinal Study on the Evolution Trend and Influencing Factors of Postoperative Reflux of Esophageal Cancer Based on PEPTEST Technique
Status: Enrolling by invitation | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: NCC4005
Record Dates: First submitted 2023-08-26; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-03

CONDITIONS: GASTROINTESTINAL NEOPLASMS
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Before surgery: A patient with esophageal cancer before surgery
  Interventions: Diagnostic Test: PEPTEST test
- Before discharge: Patients with esophageal cancer who were not discharged after surgery
  Interventions: Diagnostic Test: PEPTEST test
- 1 month after surgery: One month after surgery for esophageal cancer
  Interventions: Diagnostic Test: PEPTEST test
- 3 months after surgery: Three months after surgery for esophageal cancer
  Interventions: Diagnostic Test: PEPTEST test
- 6 months after surgery: Six months after surgery for esophageal cancer
  Interventions: Diagnostic Test: PEPTEST test

INTERVENTIONS:
Diagnostic Test: PEPTEST test — Quantitative determination of gastric salivary amylase。

SUMMARY:
The goal of this observational study intends to explore the evolution trend and related factors of postoperative reflux of esophageal cancer based on PEPTEST detection, in order to identify postoperative reflux

The main question it aims to answer are:

to provide evidence for high-risk groups, improvement of surgical methods for esophageal cancer, and development of health education programs to prevent postoperative reflux.

Using convenient sampling method, patients undergoing esophagectomy in thoracic surgery Department of Cancer Hospital of Chinese Academy of Medical Sciences from January 1, 2023 were continuously enrolled. PEPTEST was performed once before surgery, before discharge, 1 month, 3 months, and 6 months after surgery.

The incidence of pathological reflux at 5 time points before and after surgery was observed and compared (that is, both T-line and C-line were shown). The trend of pepsin content in saliva before and after operation; The relationship between pathological reflux and surgical factors; The relationship between pathological reflux and life habits after operation; Relationship between pathological regurgitation and demographic characteristics.

DETAILED DESCRIPTION:
The subjects of this study were selected from the patients who underwent esophagectomy in the Department of Thoracic Surgery of Cancer Hospital of Chinese Academy of Medical Sciences from January 1, 2023 to December 1, 2023, and the patients who underwent esophagectomy in the Department of thoracic surgery of Cancer Hospital of Chinese Academy of Medical Sciences from January 1, 2023. PEPTEST was performed once before surgery, before discharge, 1 month, 3 months, and 6 months after surgery. To describe the evolution trend of postoperative reflux in patients with esophageal cancer can be used for anticipatory sexual health education. To explore the relevant factors of reflux: to identify the inherent factors, such as gender, BMI, etc., to give preventive intervention to high-risk groups; The variable factors such as the length and width of the tube stomach can be improved.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were pathologically diagnosed with esophageal cancer and underwent esophagectomy for esophageal cancer.
2. The patient can communicate in Mandarin.
3. Those who can come to the hospital for review on time.

Exclusion Criteria:

1. People with cognitive impairment or mental illness.
2. Complicating other serious life-threatening diseases (such as leukemia or autoimmune diseases).
3. Unwilling to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent resection for esophageal cancer were continuously enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of pathological regurgitation | 2023.1.1-2023.12.1
  Incidence of pathological regurgitation at 5 time points before and after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No